CLINICAL TRIAL: NCT04701593
Title: Using Intraoperative Triamcinolone Acetonide Irrigation to Reduce Post-Operative Pain From Scleral Buckle Surgery
Brief Title: Using Triamcinolone Acetonide to Reduce Pain After Scleral Buckle Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19-377
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Retinal Detachment
Keywords: Scleral Buckle; Triamcinolone Acetonide
MeSH Terms: conditions — Retinal Detachment | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): No additional drug given
- Experimental (Triamcinolone Acetonide) (Experimental): receives a sub-tenon irrigation of 1 cc 40mg/mL triamcinolone acetonide around the base of the scleral buckle (0.25 cc in each quadrant) at time of operation
  Interventions: Drug: Triamcinolone Acetonide 40mg/mL

INTERVENTIONS:
Drug: Triamcinolone Acetonide 40mg/mL — Sub-tenon irrigation 1cc
  Other Names: Kenalog
  Arms: Experimental (Triamcinolone Acetonide)

SUMMARY:
PURPOSE: Scleral buckle surgery is a widely used ophthalmic surgery for the correction of rhegmatogenous retinal detachment. Studies suggest that eye pain is a common and underestimated occurrence after scleral buckle surgery, but as of yet, there is no definitive management method for reducing pain following scleral buckle surgery. The investigators aim to control pain following scleral buckle surgery with sub-tenon's irrigation with triamcinolone acetonide at the time of surgery. Using a randomized prospective clinical study, the investigators test if this technique will reduce the pain, nausea/vomiting, and analgesic use caused by scleral buckle surgery.

METHODS: Forty-eight patients undergoing scleral buckle surgery will be randomized into two groups. The experimental group receives a sub-tenon irrigation of 1 cc 40mg/mL triamcinolone acetonide around the base of the scleral buckle (0.25 cc in each quadrant) at time of operation. The control group does not receive any triamcinolone irrigation. Pain scores are measured 1 day post-operatively via 11-pt numerical rating scale as the primary outcome. The nausea/vomiting score is measured 1 day post-operatively via standard 6-pt scale. Patients track pain medication use via pill count. Values will be measured again at 1-2-week and 6 months post-op.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have rhegmatogenous retinal detachment and be scheduled to undergo scleral buckle surgery for correction

Exclusion Criteria:

* Advanced Glaucoma
* History of corticosteroid responsive elevation in IOP
* Allergy to Triamcinolone Acetonide or other corticosteroids
* Pre-existing chronic pain disorders
* Herpes zoster
* Prior corneal allograft
* Allergy to local anesthetic or penicillin
* Patients unable to consent on own behalf
* Patients unable to communicate pain and nausea levels
* Pregnancy
* Incarceration

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vishak J John, MD, Principal Investigator — Virginia Tech, Vistar Eye Center
Locations (1):
- Vistar Eye Centers, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Experimental (Triamcinolone Acetonide)
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental (Triamcinolone Acetonide) | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Customized [Count of Participants; unit: Participants]
  <20 years | 0 | 0 | 0
  20-40 years | 0 | 2 | 2
  40-65 years | 5 | 4 | 9
  65+ years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 9 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Pain Day 1
Description: 11-point Numerical Rating Scale (0-10, 10 being highest level of pain)
Time Frame: 1 Day Post-Op
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Experimental (Triamcinolone Acetonide)
Number analyzed (Participants) | 5 | 9
score on a scale | 2.2 [2 to 3] | 1.0 [0 to 1.75]

2. Secondary Outcome: Post Operative Pain Week 1
Description: 11-point Numerical Rating Scale (0-10, 10 being highest level of pain)
Time Frame: 1 Week Post-Op
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Experimental (Triamcinolone Acetonide)
Number analyzed (Participants) | 5 | 9
score on a scale | 0.8 [0 to 1] | 0 [0 to 0]

3. Secondary Outcome: Pain Medication Use (Tylenol in mg)
Description: Amount of Tylenol used (in mg) cumulatively over one week after the operation
Time Frame: Cumulative amount used was assessed at one week after operation
Measure: Mean (Inter-Quartile Range); unit: milligrams
Arm/Group | Control | Experimental (Triamcinolone Acetonide)
Number analyzed (Participants) | 5 | 9
milligrams | 3125 [250 to 3300] | 2403 [0 to 2500]

ADVERSE EVENTS:
Time Frame: 6 months after experimental treatment
Description: There is no risk for mortality from the use of FDA approved intraocular steroids, no such event has ever been reported
Arm/Group | Control | Experimental (Triamcinolone Acetonide)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=5) | Experimental (Triamcinolone Acetonide) (N=9)
Infection (Eye disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT04701593/Prot_SAP_000.pdf